CLINICAL TRIAL: NCT04875403
Title: Physical Functional Impacts of Rehabilitation in Patients With Human Lymphotropic Virus Type I
Brief Title: Rehabilitation in Patients With Human Lymphotropic Virus Type I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Metodista de Piracicaba (Other)
Collaborators: Universidade do Estado do Pará (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, Researcher, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01/2021
Record Dates: First submitted 2021-04-27; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Human T-Lymphotropic Virus Type 1 Associated Myelopathy
MeSH Terms: conditions — Paraparesis, Tropical Spastic | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory muscle training group (Experimental): Inspiratory muscle training with linear load device, associated with the resisted training. The initial training load for each participant will be adjusted to 25% of MIP. Each week, the researcher determines the new values for load (1 to week 25%, 2 to week 35%;. 3 to week 40%;. 4 to week 45%;. 5 to week 50%.).The resistance training protocol will consist of the exercises of the front pull, the extension chair and the vertical bench press, covering large muscle groups in the dorsal region of the quadriceps and chest, respectively. Each year consist of three sets of 10 repetitions with a load equivalent to 60% of a test Repetition Maximum (1RM), which will be changed every week (1 to week 60%, 2 to week 65%;. 3 the . week 70%, 4 to week. 75%, 5 to week 80%).
  Interventions: Other: Inspiratory muscle trainning
- Aerobic exercise group (Active Comparator): Exercise bike for 30 minutes, which will be divided into 10 minutes for the foot heating and 20 minutes for the workout aerobic exercise that will have to maintain a target training heart rate, training has to be equivalent to 40% to 60%% target intensity.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Inspiratory muscle trainning — linear load device, associated with the resisted training. The initial training load for each participant will be adjusted to 25% of MIP. Each week, the researcher determines the new values for load (1 to week 25%, 2 to week 35%;. 3 to week 40%;. 4 to week 45%;. 5 to week 50%.).
  Arms: Respiratory muscle training group
Other: Exercise — exercise bike for 30 minutes, which will be divided into 10 minutes for the foot heating and 20 minutes for the workout aerobic exercise that will have to maintain a target training heart rate
  Arms: Aerobic exercise group

SUMMARY:
In our times, it is known that approximately 5% of patients seropositive for HTLV-1 may desengage a frame with several neurological disorders, which is called myelopathy associated with HTLV-1, characterized for gait, decreased dynamic balance and limitation of walking independence the use of walkers, crutches as in wheelchairs. This evolution of the disease is based, above all, on muscle changes, such as inflammation of the muscles, which contributes to the attenuation of muscle capacity . In addition, muscle changes caused by HTLV-1 also affect the respiratory muscles, causing a change in respiratory mechanics, which can impair alveolar ventilation and, therefore, the development of a restorative respiratory disorder, reducing total lung capacity. Therefore, it is perceived the importance of offering planned rehabilitation according to the global assessment of the health status of these patients, considering their influence on activities of daily living.The focus of this study is on the weekly respiratory muscle training, as assessed by mensuration maximal inspiratory pressure, showed significant results in improving lung capacity and in this way promoting the prevention of pulmonary complications. Therefore, the protocol proposed by the present study includes respiratory muscular training plus resistance exercise, assessing the impact on both the strength muscular respiratory to as peripheral muscles, through the palmar pressure test and consequent enhancement of quality life and functionality of these patients. Furthermore, it will be possible to contribute to the knowledge of society and the scientific community about this theme, which is still very small in the world literature.

ELIGIBILITY:
Inclusion Criteria:

* Seropositive carriers for HTLV-1 with PET

Exclusion Criteria:

* lung diseases
* heart disease
* arterial hypertension
* cognitive impairments

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscular strenght | from baseline respiratory muscle stenght to 5 weeks
  The assessment of respiratory muscle strength will be carried out weekly by measuring the maximum inspiration pressure
Functional capacity | from baseline functional capacity to 5 weeks
  The assessment of functional capacity will be carried out weekly by six minute walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade do Estado do Pará, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hirons A, Khoury G, Purcell DFJ. Human T-cell lymphotropic virus type-1: a lifelong persistent infection, yet never truly silent. Lancet Infect Dis. 2021 Jan;21(1):e2-e10. doi: 10.1016/S1473-3099(20)30328-5. Epub 2020 Sep 25. PMID 32986997
- [Result] Pereira FM, Almeida MDCC, Santos FLN, Carreiro RP, Galvao-Castro B, Grassi MFR. Distribution of Human T-Lymphotropic Virus (HTLV) and Hepatitis C Co-infection in Bahia, Brazil. PLoS One. 2020 Jul 21;15(7):e0223087. doi: 10.1371/journal.pone.0223087. eCollection 2020. PMID 32692782